CLINICAL TRIAL: NCT05949424
Title: Optimal Dosing of Oral Anticancer Drugs in Older Adults With Cancer: a Randomized Pilot Study.
Brief Title: OPTI - DOSE: Optimal Dosing of Oral Anticancer Drugs in Older Adults
Acronym: OPTI-DOSE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16800
Record Dates: First submitted 2023-06-19; First posted 2023-07-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Renal Cell Carcinoma; Ovarian Carcinoma; Thyroid Carcinoma; Breast Carcinoma; Endometrium Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Ovarian Neoplasms; Thyroid Neoplasms; Breast Neoplasms; Endometrial Neoplasms | interventions — olaparib; lenvatinib; Sunitinib; palbociclib; pazopanib

STUDY DESIGN:
Intervention Model Description: Control group: standard SmPC dosing. Intervention group: lower starting dose with dose-escalation inversely following the dosing steps from the SmPC every 2 weeks in case of good tolerability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Standard SmPC dosing with dose adjustments for toxicity as per SmPC
  Interventions: Drug: Olaparib; Drug: Lenvatinib; Drug: Sunitinib; Drug: Palbociclib; Drug: Pazopanib
- Intervention group (Experimental): Lower starting dose with dose-escalation inversely following the dosing steps from the SmPC every 2 weeks in case of good tolerability
  Interventions: Drug: Olaparib; Drug: Lenvatinib; Drug: Sunitinib; Drug: Palbociclib; Drug: Pazopanib

INTERVENTIONS:
Drug: Olaparib — Starting dose of 200mg 2dd.
  Other Names: Lynparza
  Arms: Intervention group
Drug: Lenvatinib — Starting dose of 10mg 1dd.
  Other Names: Lenvima
  Arms: Intervention group
Drug: Sunitinib — Starting dose of 25mg 1dd 28/42 days.
  Other Names: Sutent
  Arms: Intervention group
Drug: Palbociclib — Starting dose of 75mg 1dd 21/28 days.
  Other Names: Ibrance
  Arms: Intervention group
Drug: Pazopanib — Starting dose of 200mg 1dd.
  Other Names: Votrient
  Arms: Intervention group
Drug: Olaparib — Starting dose of 300mg 2dd.
  Other Names: Lynparza
  Arms: Control group
Drug: Lenvatinib — Starting dose of 20mg 1dd for RCC or endometrial carcinoma, starting dose of 24mg 1dd for thyroid carcinoma.
  Other Names: Lenvima
  Arms: Control group
Drug: Sunitinib — Starting dose of 50mg 1dd 28/42 days.
  Other Names: Sutent
  Arms: Control group
Drug: Palbociclib — Starting dose of 125mg 1dd 21/28 days.
  Other Names: Ibrance
  Arms: Control group
Drug: Pazopanib — Starting dose of 800mg 1dd.
  Other Names: Votrient
  Arms: Control group

SUMMARY:
The study hypothesis is that a lower starting dose of anticancer tablet treatments can lead to better treatment tolerability in older patients, while the benefits of treatment can be the same. The trial population consists of 30 patients aged 65 years or older, who are starting treatment with one of these anti cancer tablet treatments: pazopanib, olaparib, lenvatinib, sunitinib or palbociclib. The control group (half of the participants) will be treated with the standard-of-care, the interventional group will start with the lowest dose of the anti cancer tablets as described in the drug label. The dose will be increased every two weeks in case of good tolerability. Results of this pilot study will be used to inform the design of the larger randomised phase 2 trial.

DETAILED DESCRIPTION:
Information about the benefits and side effects of treatments for cancer is mainly derived from studies with younger patients. It is known that elderly patients experience more side effects from treatments, which can lead to a worse quality of life. The study hypothesis is that a lower starting dose of anticancer tablet treatments can lead to better treatment tolerability in older patients, while the benefits of treatment can be the same.

The trial population consists of 30 patients aged 65 years or older, who are starting treatment with one of these anti cancer tablet treatments: pazopanib, olaparib, lenvatinib, sunitinib or palbociclib. This is a randomized study with 1:1 randomisation, stratified by type of anti-cancer treatment.

The control group (half of the participants) will be treated with the standard-of-care, that means with the recommended starting dose of the anti cancer tablets as described in the drug label. The dose can be adjusted (lowered) if this is necessary, for example because of side effects, based on the judgment of the treating physician. The interventional group (half of the participants) will start with the lowest dose of the anti cancer tablets as described in the drug label. The dose will be increased every two weeks in case of good tolerability. Results of this pilot study will be used to inform the design of the larger randomised phase 2 trial, for example the primary endpoint, the amount of investigations and the size of the study population.

Study visits are planned every 2 weeks for a total study duration of 12 weeks, the time point for analysis of the primary endpoint. Blood samples for PK analysis are collected every 2 weeks. A baseline blood sample will be collected for pharmacogenomic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 65 years of age.
* Indication for starting treatment with pazopanib (for renal cell carcinoma), olaparib (for ovarian carcinoma), lenvatinib (as monotherapy for thyroid carcinoma, or in combination with pembrolizumab for renal cell carcinoma or endometrium carcinoma), sunitinib (for renal cell carcinoma) or palbociclib (for breast carcinoma).
* No contra-indications for starting treatment at the recommended starting dose as per SmPC.
* All patients must provide written informed consent prior to enrolment.

Exclusion Criteria:

• Planned starting dose lower than the recommended starting dose as per SmPC

For Pazopanib:

* Use of a strong CYP3A4-inhibitor or PgP-inhibitor
* Creatinine clearance <30ml/min
* Moderate or severe hepatic impairment (bilirubin >1.5x ULN)

For Olaparib:

* Use of a moderate or strong CYP3A4-inhibitor
* Creatinine clearance <50 ml/min
* Severe hepatic impairment (Child-Pugh 10-15)

For Lenvatinib:

* Creatinine clearance <30ml/min
* Severe hepatic impairment (Child-Pugh score 10-15)

For Sunitinib:

* Use of a strong CYP3A4-inhibitor
* Use of a strong CYP3A4-inducer

For Palbociclib:

* Use of a strong CYP3A4-inhibitor
* Severe hepatic impairment (Child-Pugh score 10-15)
* Other findings at interview or physical examination that hamper compliance to the study protocol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of investigating whether a lower starting dose with step-up approach leads to a better overall treatment utility compared to standard dosing | 12 weeks
  * The percentage of patients that are willing to participate, from all eligible patients
  * The percentage of patients that successfully complete the first 12 weeks of the trial
  * The percentage of data points that are successfully collected during the first 12 weeks of the trial

SECONDARY OUTCOMES:
Overall treatment utility | 12 weeks
  measured by the investigator. See: https://blogs.ed.ac.uk/canceroutcomes/overall-treatment-utility/#:~:text=In%20Oncology%20clinical%20research%2C%20Overall%20Treatment%20Utility%20%28OTU%29,balance%20of%20benefits%20and%20harms%20from%20cancer%20treatments
Progression free survival | up to 60 months
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Overall survival | up to 60 months
  From date of randomization until the date of death from any cause, assessed up to 60 months
Quality of life | 12 weeks
  measured by QLQ-C30 (general) and QLQ-ELD14 (elderly cancer patients)
Safety | 12 weeks
  Adverse events, measured by CTCAE v5.0
Hospital care use | 12 weeks
  number of outpatients visits, telephone contacts or hospital admission days
Pharmacokinetic parameters: Cmax | 12 weeks
  Peak Plasma Concentration (Cmax)
Pharmacokinetic parameters: AUC | 12 weeks
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetic parameters: Ctrough | 12 weeks
  Trough Plasma Concentration (Ctrough)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Broekman, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided